CLINICAL TRIAL: NCT02505659
Title: Efficacy of Preoperative Re-education on Patients With an Anterior Cruciate Ligament Rupture: a Randomized Controlled Trial
Brief Title: Efficacy of Preoperative Re-education on Patients With an Anterior Cruciate Ligament Rupture
Acronym: PRELIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0240; 2014-A01845 (Registry Identifier: 2014-A01845-42)
Record Dates: First submitted 2015-06-26; First posted 2015-07-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament rupture; Preoperative re-education; Knee functional performance; Anterior cruciate ligament surgery; Single-leg hop for distance test performance
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Sessions are aiming to neuromuscular and functional training. Each session starts with trunk muscle activation. Patients will then have to realize a neuromuscular training on Huber Motion Lab® followed by multiple exercises targeting functional stability and neuromuscular control. From the 4th session, a jump sequence will be added to the previous exercices. Exercises used in this protocol are based upon successful exercises of protocols already performed on patients with anterior cruciate ligament rupture.
  Interventions: Behavioral: Preoperative re-education
- CONTRL GROUP (No Intervention): a control group (without preoperative reeducation)

INTERVENTIONS:
Behavioral: Preoperative re-education — Preoperative re-education (behavior): 8 re-education sessions of 30 to 40 minutes, 2 times a week, for 4 weeks
  Arms: EXPERIMENTAL GROUP

SUMMARY:
Anterior cruciate ligament (ACR) rupture is a common lesion of sportsmen that leads to functional deficits which are difficult to overcome. To prevent from an unfavorable evolution, patients can either get a non-surgical treatment or an ACR surgery, which is very common. Knee functional performance level could impact on the postoperative outcome and it's of common knowledge that early re-education after an ACR rupture improves knee functioning.

Patients with an ACR rupture enrolled in this study will be randomized either in an experimental group (with preoperative reeducation) or in a control group (without preoperative reeducation). Both groups will then have post-operative re-education (40 sessions) based on HAS recommendations.

The main aim of this study is to assess the impact of preoperative re-education on knee functional performance 4 month after surgical reconstruction of an ACR.

Secondary aims are to determine the impact of the 4-week preoperative re-education on knee functional performance after an ACR rupture, before surgery and 7 months after surgery.

Functional performance, muscular strength, proprioception and anterior knee laxity will be measured at inclusion (V0), 4-5 days before surgery (V1), 4 month (V4M) and 7 months (V7M) after surgery. Lysholme-Tegner scoring and IKDC2000 questionnaire will be added to the previous assessments.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACR) rupture is a common lesion of sportsmen that leads to functional deficits which are difficult to overcome. To prevent from an unfavorable evolution, patients can either get a non-surgical treatment or an ACR surgery, which is very common. Knee functional performance level could impact on the postoperative outcome and it's of common knowledge that early re-education after an ACR rupture improves knee functioning.

Patients with an ACR rupture enrolled in this study will be randomized either in an experimental group (with preoperative reeducation) or in a control group (without preoperative reeducation). Both groups will then have post-operative re-education (40 sessions) based on HAS recommendations.

The main aim of this study is to assess the impact of preoperative re-education on knee functional performance 4 month after surgical reconstruction of an ACR.

Secondary aims are to determine the impact of the 4-week preoperative re-education on knee functional performance after an ACR rupture, before surgery and 7 months after surgery.

Functional performance, muscular strength, proprioception and anterior knee laxity will be measured at inclusion (V0), 4-5 days before surgery (V1), 4 month (V4M) and 7 months (V7M) after surgery. Lysholme-Tegner scoring and IKDC2000 questionnaire will be added to the previous assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 45 years old
* Tegner physical activity level between 3 and 9
* Primary and unilateral rupture of anterior cruciate ligament, confirmed by MRI
* patient available to carry out the preoperative re-education program

Exclusion Criteria:

* Complex lesion that would impede on preoperative re-education (posterior cruciate ligament, meniscal or chondral symptomatic lesion, fracture)/
* Neurologic or cardiorespiratory pathology contra-indicating preoperative re-education
* Previous surgical treatment of the lower limbs or of the lumbar spine
* Neuropathic or algodystrophic pain on the lower limbs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Functional performance as assessed by single-leg hop for distance test performance | at 4 months after ACR surgery.

SECONDARY OUTCOMES:
Ability to return to high level athletics as assessed by single-leg hop for distance test performance | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for:
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Dynamic balance as assessed by star excursion balance test | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for:
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Quadriceps muscular strength as assessed by isokinetic test of quadriceps muscular strength | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for:
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Proprioception as assessed by repositioning knee test | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for:
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Knee anterior stability as assessed by KT-1000 | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Subjective knee evaluation as assessed by International Knee Documentation committee 2000 questionnaire | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Knee symptoms as assessed by Lysholme questionnaire | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)
Physical activity level as assessed by Tegner knee scoring | at 4-month follow-up and 7-month follow-up compared to the initial visit and control group for
  Assessment for both control and experimental group : inclusion (V0) preoperative visit (V1), 4-month follow-up (V4M) and 7-month follow-up (V7M)

CONTACTS AND LOCATIONS:
Overall Officials: Aurore CHABAUD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France